CLINICAL TRIAL: NCT05593198
Title: Randomized Controlled Clinical Trial Comparing the Clinical Measures and the Radiographical Volumetric Outcomes Assessed by Cone Beam Computed Tomography of Guided Bone Regeneration Versus Bone Block Grafting
Brief Title: Guided Bone Regeneration Versus Bone Block Grafting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 4729
Record Dates: First submitted 2022-09-05; First posted 2022-10-25 (Actual); Last update posted 2023-08-29 (Actual); Status verified 2022-10

CONDITIONS: Atrophy; Bone
Keywords: Bone Regeneration
MeSH Terms: conditions — Atrophy

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Guided bone regeneration (Active Comparator): Patients will be treated with guided bone regeneration.
  Interventions: Procedure: Guided bone regeneration
- Bone block (Experimental): Patients will be treated with bone blocks using the Khoury technique.
  Interventions: Procedure: Khoury technique

INTERVENTIONS:
Procedure: Khoury technique — the bone block will be used following the principles of the Khoury technique to augment the bone volume.
  Arms: Bone block
Procedure: Guided bone regeneration — the membrane and the bone granules will be used to perform the guided bone regeneration technique.
  Arms: Guided bone regeneration

SUMMARY:
The purpose of this study is to analyze the volumetric gain and stability of the newly formed bone tissue comparing guided bone regeneration with block graft.

ELIGIBILITY:
Inclusion Criteria:

* Patients in need of an implant-supported rehabilitation
* Patients requiring bone regeneration
* Healthy patients
* Full-mouth plaque score (FMPS) and full-mouth bleeding score (FMBS) ≤ 15%
* Sufficient mesiodistal and interocclusal space
* At least 6 months of follow-up

Exclusion Criteria:

* An American Society of Anesthesiologists physical status classification ≥ III
* General contraindications for surgical treatment or implant placement
* Untreated periodontitis
* Smoking
* Excessive alcohol consumption
* Any drug or medication known to affect oral status and bone turnover or contraindicate surgical treatment
* No residual keratinized tissue at the experimental area
* Unwillingness to return for follow-up examinations

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2023-07-01 (Actual); Study Completion 2023-07-02 (Actual)

PRIMARY OUTCOMES:
Bone volume | 6 Months follow up
  the bone volume will be analyzed with the Cone Beam Computed Tomography scan

SECONDARY OUTCOMES:
Periodontal parameters | 6 Months follow up
  the periodontal parameters will be analyzed clinically with the periodontal probe and measured in millimeters. All the periodontal parameters will be combined to describe the periodontal status of the patient.
Wound healing | 2 weeks follow up
  the wound healing will be recorded with the Early Wound Healing Score (EHS) ranging from 0 to 10 which includes the following parameters:
  * clinical signs of re-epithelialization: 0 points, visible distance between incision margins; 3 points, incision margins in contact; 6 points, merged incision margins.
  * clinical signs of haemostasis: 0 points, bleeding at the incision margins; 1 point, presence of fibrin at the incision margins; 2 points, absence of fibrin on the incision margins.
  * clinical signs of inflammation: 0 points, redness involving >50% of the incision length and/or pronounced swelling; 1 point, redness involving <50% of the incision length; 2 points, absence of redness along the incision length.
Histological analysis | 6 Months follow up
  The histological analysis will be performed harvesting a sample during the implant placement. Bone biopsies including both native and regenerated bone will be subjected to digital scanning to analyze the characteristics of newly formed bone, the remaining grafted material, integration of grafted material with newly formed bone, soft tissue, and local inflammation. Histomorphometric analyses will be performed to measure the following parameters: bone tissue area , graft material area , soft tissue area. Bone tissue area , graft material area , soft tissue area will be expressed relative to the total area.

CONTACTS AND LOCATIONS:
Overall Officials: Antonio D'Addona, DDS, Principal Investigator — Fondazione Policlinico Gemelli
Locations (1):
- Fondazione Policlinico Gemelli, Rome, Italy

IPD SHARING:
Plan to Share IPD: No